CLINICAL TRIAL: NCT01789736
Title: A Study Assessing the Safety and Ocular Hypotensive Efficacy of PG286 Ophthalmic Solution, 0.5% Compared to Its Individual Components
Brief Title: A Study Assessing PG286 Ophthalmic Solution, 0.5% Compared to Its Individual Components for 28 Days
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PG286-CS202
Record Dates: First submitted 2013-02-09; First posted 2013-02-12 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular hypertension; AR-12286; Travoprost
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PG286 (Experimental): PG286 Ophthalmic Solution q.d. O.U.
  Interventions: Drug: PG286 Ophthalmic Solution 0.5%
- AR-12286 Ophthalmic Solution 0.5% (Experimental): AR-12286 Ophthalmic Solution 0.5% q.d. O.U.
  Interventions: Drug: AR-12286 Ophthalmic Solution 0.5%
- Travoprost 0.004% (Active Comparator): Travoprost 0.004% q.d. O.U.
  Interventions: Drug: Travoprost Ophthalmic Solution 0.004%

INTERVENTIONS:
Drug: PG286 Ophthalmic Solution 0.5% — PG286 Ophthalmic Solution
  Arms: PG286
Drug: AR-12286 Ophthalmic Solution 0.5% — AR-12286 Ophthalmic Solution 0.5%
  Arms: AR-12286 Ophthalmic Solution 0.5%
Drug: Travoprost Ophthalmic Solution 0.004% — Travoprost Ophthalmic Solution 0.004%
  Arms: Travoprost 0.004%

SUMMARY:
In the double-masked, randomized, multi-center, active-controlled parallel study, patients will be randomized to receive either a fixed dose combination of AR-12286 and travoprost, AR-12286, or travoprost. The hypothesis is that there is no difference between each treatment arm.

ELIGIBILITY:
Subject inclusion criteria

1. 18 years of age or greater.
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
3. Unmedicated (post-washout) IOP ≥ 22 mm Hg at 2 qualification visits (08:00 hr), 2-7 days apart. At second qualification visit, IOP >21 mmHg at 10:00 and 16:00 hrs.
4. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
5. Able and willing to give signed informed consent and follow study instructions.

Subject exclusion criteria

Excluded from the study will be individuals with the following characteristics:

Ophthalmic (in either eye):

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure, or narrow angles. Note: Previous laser peripheral iridotomy is NOT acceptable.
2. Intraocular pressure > 35 mm Hg, or use of more than two ocular hypotensive medications within 30 days of screening. Note: fixed dose combinations count as two medications.
3. Known hypersensitivity to any component of the formulation (benzalkonium chloride, zinc, etc.), travoprost, or to topical anesthetics.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s).
5. Refractive surgery in study eye(s) (e.g., radial keratotomy, PRK, LASIK, etc.).
6. Ocular trauma within the six months prior to screening, or ocular surgery or laser treatment within the three months prior to screening.
7. Evidence of ocular infection, inflammation, clinically significant blepharitis, conjunctivitis, or a history of herpes simplex keratitis at screening.
8. Ocular medication of any kind within 30 days of screening, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after screening) or c) lubricating drops for dry eye (which may be used throughout the study).
9. Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (e.g., cup-disc ratio > 0.8).
10. Central corneal thickness greater than 600 µm.
11. Any abnormality preventing reliable applanation tonometry of either eye.

    Systemic:
12. Clinically significant abnormalities (as determined by the investigator) in laboratory tests at screening.
13. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
14. Participation in any investigational study within 30 days prior to screening.
15. Changes of systemic medication within 30 days prior to screening, or anticipated during the study, that could have a substantial effect on IOP.
16. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mean diurnal IOP | 28 Days
  The primary efficacy endpoint will be the mean diurnal IOP across subjects within treatment group and time point at Day 28.

SECONDARY OUTCOMES:
IOP | 7-28 days
  Secondary efficacy endpoints will include: mean IOP across subjects within treatment group at each post-treatment timepoint, mean change from diurnally adjusted baseline IOP at each timepoint, mean percent change from diurnally adjusted baseline IOP at each timepoint, mean diurnal IOP at other visits, and mean change from the baseline mean diurnal IOP at each visits.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Kenneth Sall, M.D., Artesia, California
  - United Medical Research Institute, Inglewood, California
  - Aesthetic Eye Care Institute, Newport Beach, California
  - Bacharach practice, Petaluma, California
  - Centre For Health Care, Poway, California
  - Clayton Eye Center, Morrow, Georgia
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Bradley Kwapiszeski, MD, Shawnee Mission, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Alan L Robin, M.D., Baltimore, Maryland
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Rochester Ophthalmological Group, Rochester, New York
  - Jeffrey Schultz, M.D., The Bronx, New York
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Belmont, North Carolina
  - The Eye Institute, Tulsa, Oklahoma
  - Texan Eye, Austin, Texas
  - Medical Center Ophth. Associates, San Antonio, Texas
  - Stacy R. Smith, M.D., Salt Lake City, Utah
  - Virginia Eye Consultants, Norfolk, Virginia